CLINICAL TRIAL: NCT04428320
Title: The Effect of Preemptive Levator Ani Injections on Pain After Pelvic Reconstructive Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-124
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Pelvic Floor Prolapse; Surgery; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivicaine pelvic floor muscle injection (Experimental): Five injections at pre-specified locations at pelvic floor muscle bilaterally after induction of general anesthesia for vaginal pelvic prolapse surgery
  Interventions: Procedure: Pelvic floor injection
- Standard of care (no injection) preoperatively (No Intervention): No injection - standard analgesia

INTERVENTIONS:
Procedure: Pelvic floor injection — Injection of 10 cc of bupivacaine
  Arms: Bupivicaine pelvic floor muscle injection

SUMMARY:
Patients undergoing vaginal pelvic reconstructive surgery for pelvic organ prolapse (POP) under general anesthesia will be randomized to receive bilateral trans-vaginal pelvic floor muscle injections with bupivacaine or no injection (standard of care) as a part of their surgical pain control

DETAILED DESCRIPTION:
Patients undergoing vaginal pelvic reconstructive surgery for pelvic organ prolapse (POP) under general anesthesia will be randomized to receive:

1. Bilateral trans- vaginal pelvic floor levator ani muscle injections (trigger point injections) with bupivacaine:

   - 0.5% bupivacaine will be injected at several sites for a total of 5ml on each side of the pelvic floor, with each injection site no more than 1 ml (Bupivacaine was chosen by the study team because of it has a longer half life then other common local anesthetics. We plan to use the same anesthetic and dosage to standardize the protocol between patients. Other local anesthetics will not be used in addition to the bupivacaine administered for research purposes. We will limit the amount of intravenous lidocaine to less than 5mg/ kg).
2. Control- No additional treatment (standard of care).

The patient will be blinded to their randomization (single blind). The post-operative pain regimen will be standardized when possible. Patients will receive a regimen of IV and oral narcotics and Ketorolac per our routine post-operative protocol. On discharge from the hospital, patients will be given prescriptions for a standard amount of oral narcotic, 20 tablets of oxycodone (150 morphine equivalents), and 30 tablets of 600mg ibuprofen.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Able to read English and give informed consent
* Undergoing VAGINAL pelvic reconstructive surgery for POP

Exclusion Criteria:

* Hypersensitivity or allergy to amide anesthetics
* Documented chronic pain condition

  o (back pain, pelvic pain, fibromyalgia, etc.)
* Bleeding disorder
* Connective tissue disorder
* Neuromuscular disorder
* Cardiac conduction abnormality or channelopathy
* Hepatic Impairment
* Renal Impairment
* History of, or current, narcotic or alcohol dependence
* History of pelvic radiation or gynecologic malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pelvic organ prolapse surgery for female genitalia
Enrollment: 140 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2022-05-21 (Estimated); Study Completion 2022-05-21 (Estimated)

PRIMARY OUTCOMES:
VAS analog scale on post-op day #1 | postop day #1

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper Health University, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
No sharing planned as of now